CLINICAL TRIAL: NCT01204918
Title: Efficacy and Tolerability of Riluzole in Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0903004917; 137889 (Other: Other); NCT01298427 (obsolete NCT alias)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Depression
Keywords: MDD; Depression; Treatment refractory; Glutamate; Riluzole; Major depressive disorder; psychopharmacology; rilutek
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Riluzole addition to SSRI antidepressant (Experimental): Riluzole 100mg added to ongoing SSRI or SNRI antidepressant for 8 weeks
  Interventions: Drug: Riluzole
- Placebo addition to standard SSRI antidepressant (Placebo Comparator): Placebo will be added to ongoing SSRI or SNRI antidepressant treatment for 8 weeks
  Interventions: Drug: placebo
- Riluzole/Placebo addition to SSRI antidepressant (Experimental): Riluzole 100mg added to ongoing SSRI or SNRI antidepressant for 4 weeks and placebo will added to ongoing SSRI or SNRI antidepressant treatment for 4 weeks
  Interventions: Drug: Riluzole; Drug: placebo

INTERVENTIONS:
Drug: Riluzole — Riluzole 100mg PO
  Other Names: Rilutek
  Arms: Riluzole addition to SSRI antidepressant; Riluzole/Placebo addition to SSRI antidepressant
Drug: placebo — placebo
  Arms: Placebo addition to standard SSRI antidepressant; Riluzole/Placebo addition to SSRI antidepressant

SUMMARY:
This study aims to examine the antidepressant efficacy of riluzole, employing a randomized, double-blind, placebo-controlled, adjunctive trial in treatment-resistant major depressive disorder (TRD).

DETAILED DESCRIPTION:
This study aims to examine the antidepressant efficacy of riluzole, employing a randomized, double-blind, placebo-controlled, 8 week trial of adjunctive trial in treatment-resistant major depressive disorder (TRD). Preclinical studies have shown riluzole to modulate Glu release and clearance, and to have potent neuroprotective properties, promoting neuro-resiliency. Other preclinical data now also show the drug to have antidepressant-like effects in rodent models used to screen for antidepressant activity. In addition, several small open-label clinical studies further suggest riluzole has antidepressant and anxiolytic properties, even in patients who do not respond to standard monoaminergic antidepressant and anxiolytic medications.

ELIGIBILITY:
Group A inclusion/exclusion

Inclusion Criteria:

1. Age 18-65
2. Written informed consent
3. Meets DSM-IV criteria (by Structured Clinical Interview for DSM-IV - SCID-I/P) for MDD, current
4. Inventory of Depressive Symptomatology - Self-Rated (IDS-SR30) score of > 20 at screening, baseline and start of double-blind phase (Phase 2)
5. May have a history of failure to respond to up to two FDA-approved antidepressants at adequate doses during the current episode for at least 8 weeks, and for inclusion into the Phase 2 subjects must have failed the 8-week prospective citalopram treatment.
6. Montgomery Asberg Depression Rating Scale (MADRS) score of 18 or higher at baseline and start of Phase 2.

Exclusion Criteria:

1. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
2. Patients who no longer meet DSM-IV criteria for MDD during the baseline visit
3. Patients who demonstrate > 50% decrease in depressive symptoms as reflected by the IDS-SR total score from screen to baseline
4. Serious suicide or homicide risk, as assessed by evaluating clinician A serious suicide risk will be considered an inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death.
5. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
6. The following DSM-IV diagnoses: substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past)
7. History of a seizure disorder or clinical evidence of untreated hypothyroidism
8. Patients requiring excluded medications (see Table 3 for details)
9. Psychotic features in the current episode or a history of psychotic features, as assessed by SCID
10. Any investigational psychotropic drug within the last 3 months
11. Have failed 3 or more adequate antidepressant trials during the current Major Depressive Episode by MGH-ATRQ criteria.
12. Patients with a history of antidepressant-induced hypomania.
13. Patients with any evidence of clinically significant liver abnormalities, or any liver transaminase level >1.5 X ULN at initial screening, or >5 x ULN during Phase 2 treatment.
14. Axis II personality disorders that are the primary purpose of treatment, or would interfere with a patient's safety or compliance.
15. Patients currently being treated for a respiratory disorder (including asthma or COPD)
16. Any subject who scores a 5 or higher on item #10 of the MADRS

Group B inclusion/exclusion

Inclusion criteria:

1. Age 18-65
2. Written informed consent
3. Meets DSM-IV criteria (by Structured Clinical Interview for DSM-IV - SCID-I/P) for MDD, current
4. Inventory of Depressive Symptomatology - Self-Rated (IDS-SR30) score of > 20 at screening and baseline visits, that is at the start of Phase 2
5. Has a history of failure to respond to 1, 2, or 3 FDA-approved antidepressants at adequate doses during the current episode for at least 8 weeks, as defined by the MGH Antidepressant Treatment Response Questionnaire (MGH-ATRQ), and must be currently on the failed SSRI for at least 8 weeks and on a stable dose for at least 4 weeks.
6. Montgomery Asberg Depression Rating Scale (MADRS) score of 18 or higher at baseline and start of Phase 2.

Exclusion Criteria

1. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
2. Patients who no longer meet DSM-IV criteria for MDD during the baseline visit
3. Serious suicide or homicide risk, as assessed by evaluating clinician A serious suicide risk will be considered an inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death.
4. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
5. The following DSM-IV diagnoses: substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past)
6. History of a seizure disorder or clinical evidence of untreated hypothyroidism;
7. Patients requiring excluded medications (see Table 3 for details)
8. Psychotic features in the current episode or a history of psychotic features, as assessed by SCID
9. Any investigational psychotropic drug within the last 3 months
10. Have failed 3 or more adequate antidepressant trials during the current Major Depressive Episode by MGH-ATRQ criteria.
11. Patients with a history of antidepressant-induced hypomania.
12. Patients with any evidence of clinically significant liver abnormalities, or any liver transaminase level >2 X ULN at initial screening, or >5 x ULN during Phase 2 treatment.
13. Axis II personality disorders that are the primary purpose of treatment, or would interfere with a patients safety or compliance.
14. Patients currently being treated for a respiratory disorder (including asthma or COPD)
15. Any subject who scores a 5 or higher on item #10 of the MADRS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Sanacora, MD PhD, Principal Investigator — Yale University; Maurizio Fava, MD, Principal Investigator — Massachusettes General Hospital; Sanjay Matthew, MD, Principal Investigator — Baylor College of Medicine; Carlos Zarate, MD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (3):
- United States (3):
  - Yale University, Yale Depression Research Program, New Haven, Connecticut
  - Massachussettes General Hospital, Depression Clinical and Research Center, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Sanacora G, Kendell SF, Levin Y, Simen AA, Fenton LR, Coric V, Krystal JH. Preliminary evidence of riluzole efficacy in antidepressant-treated patients with residual depressive symptoms. Biol Psychiatry. 2007 Mar 15;61(6):822-5. doi: 10.1016/j.biopsych.2006.08.037. Epub 2006 Dec 4. PMID 17141740
- [Background] Zarate CA Jr, Payne JL, Quiroz J, Sporn J, Denicoff KK, Luckenbaugh D, Charney DS, Manji HK. An open-label trial of riluzole in patients with treatment-resistant major depression. Am J Psychiatry. 2004 Jan;161(1):171-4. doi: 10.1176/appi.ajp.161.1.171. PMID 14702270
- [Derived] Kheirkhah M, Hejazi NS, Nugent AC, Gilbert JR, Leistritz L, Walter M, Duncan WC Jr, Goldman D, Zarate CA Jr. Exploring the link between waking gamma and sleep delta power in healthy volunteers and individuals with treatment-resistant depression. J Affect Disord. 2025 Sep 15;385:119448. doi: 10.1016/j.jad.2025.119448. Epub 2025 May 19. PMID 40398609
- [Derived] Kheirkhah M, Duncan WC Jr, Yuan Q, Wang PR, Jamalabadi H, Leistritz L, Walter M, Goldman D, Zarate CA Jr, Hejazi NS. REM density predicts rapid antidepressant response to ketamine in individuals with treatment-resistant depression. Neuropsychopharmacology. 2025 May;50(6):941-946. doi: 10.1038/s41386-025-02066-7. Epub 2025 Feb 15. PMID 39955416
- [Derived] Hejazi NS, Farmer CA, Oppenheimer M, Falodun TB, Park LT, Duncan WC Jr, Zarate CA Jr. The relationship between the HDRS insomnia items and polysomnographic (PSG) measures in individuals with treatment-resistant depression. J Psychiatr Res. 2022 Apr;148:27-33. doi: 10.1016/j.jpsychires.2022.01.022. Epub 2022 Jan 11. PMID 35092868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
Started | 25 | 39 | 40
Stage 1 Begin | 25 | 39 | 40
Stage 1 End | 22 | 35 | 36
Stage 2 Begin | 22 | 35 | 36
Stage 2 End | 21 | 29 | 35
Completed | 21 | 29 | 35
Not Completed | 4 | 10 | 5
Not completed — Withdrawal by Subject | 4 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant | Total
Number analyzed (Participants) | 25 | 39 | 40 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (12.7) | 47.3 (12.1) | 46.3 (12.7) | 46.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 24 | 21 | 54
  Male | 16 | 15 | 19 | 50
Antidepressant (Y/N) [Count of Participants; unit: Participants]
  Yes | 16 | 25 | 24 | 65
  No | 9 | 14 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery and Asberg Depression Rating Scale (MADRS)
Description: This 10 item instrument is completed by the clinician by using a structured interview and defined anchor points, and aims to quantify the degree of depression over the past 7 days. The MADRS is a widely studied instrument for depression, and its reliability and validity are high. This instrument is administered at every study visit during the double-blind RCT, and at the screening, and baseline. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Usual cutoff points are:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: 4 weeks of therapy (baseline to week 4)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
Number analyzed (Participants) | 25 | 39 | 40
units on a scale | 3.20 (3.86) | 5.77 (0.52) | 4.83 (7.85)

2. Primary Outcome: Change in Montgomery and Asberg Depression Rating Scale (MADRS)
Description: as for outcome 1
Time Frame: 4 weeks of therapy (week 4 to week 8)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
Number analyzed (Participants) | 25 | 39 | 40
units on a scale | 4.13 (6.82) | 0.84 (5.79) | 3.87 (6.49)

3. Secondary Outcome: Responders Having at Least a 50% Improvement in MADRS Compared to the Baseline
Description: Responders having at least a 50% improvement in MADRS compared to the baseline in the sequential parallel design
Time Frame: 8 weeks therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
Number analyzed (Participants) | 25 | 39 | 40
Participants | 6 | 8 | 10

4. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE-SI)
Description: A commonly used instrument originally developed by NIMH and adapted into a self-report instrument. The version of the scale that we plan to use examines in a systematic fashion all possible treatment-emergent side effects and probes specific adverse symptoms, including suicidal thoughts and behaviors, and self-injurious behavior. Presented below are counts of people that had experienced the event by 8 weeks.
Time Frame: 8 weeks
Population: All subjects are included in the analysis- with the exception of sex specific conditions.
Measure: Number; unit: participants
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
Number analyzed (Participants) | 25 | 39 | 40
participants
  Trouble Sleeping | 17 | 24 | 21
  Nightmares | 9 | 15 | 11
  Drowsy | 14 | 25 | 22
  Nervousness | 13 | 19 | 14
  Fatigue | 14 | 26 | 28
  Irratibility | 15 | 22 | 23
  Poor Memory | 16 | 23 | 24
  Poor Concentration | 16 | 28 | 25
  Strange Feeling/Unreal | 4 | 7 | 5
  Hearing/Seeing Things | 1 | 2 | 1
  Abnormal Sensation | 3 | 5 | 3
  Numbness/Tingling | 2 | 8 | 4
  Dizziness | 7 | 10 | 4
  Headache | 8 | 14 | 13
  Blurred Vision | 5 | 8 | 5
  Ringing Ears | 4 | 9 | 8
  Stuffy Nose | 5 | 14 | 10
  Dry mouth | 3 | 10 | 10
  Drooling/Salivation | 2 | 4 | 0
  Muscle Cramp | 5 | 16 | 12
  Muscle Twitch | 7 | 10 | 6
  Trouble Sitting | 9 | 16 | 14
  Tremors/Shakiness | 8 | 9 | 6
  Poor Coordination | 6 | 11 | 5
  Slurred Speech | 1 | 5 | 3
  Rapid Heartbeat | 8 | 13 | 9
  Hyperventilation | 6 | 7 | 3
  Chest Pain | 4 | 6 | 2
  Nausea/Vomiting | 3 | 5 | 3
  Stomach Discomfort | 5 | 12 | 9
  Constipation | 3 | 5 | 10
  Diarrhea | 2 | 7 | 11
  Difficulty Urinating | 4 | 6 | 1
  Frequent Urination | 7 | 10 | 6
  Menstrual Irregularities: number analyzed (Participants) | 9 | 24 | 21
  Menstrual Irregularities | 0 | 2 | 1
  Loss of Sexual Interest | 13 | 26 | 22
  Sexual Performance Problems | 12 | 20 | 16
  Delayed/Absent Orgasm | 9 | 19 | 16
  Sweating Excessively | 9 | 10 | 14
  Fluid Retention | 4 | 6 | 8
  Decreased Appetite | 5 | 7 | 8
  Increased Appetite | 8 | 8 | 15
  Weight Gain | 7 | 8 | 15
  Weight Loss | 5 | 7 | 7
  Skin Rash | 3 | 4 | 3
  Diminished Mental Acuity | 16 | 22 | 22
  Difficulty Finding Words | 15 | 21 | 18
  Apathy Emotional Indifference | 11 | 18 | 21
  Dizzy When Standing Up | 8 | 10 | 2
  Bruising | 4 | 2 | 2
  Hair Thinning | 2 | 6 | 8
  Hot Flashes | 2 | 7 | 12
  Clenching Teeth | 4 | 13 | 7
  Strange Taste in Mouth | 3 | 8 | 5
  Unable to Sit Still | 9 | 17 | 14

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: These are events that were deemed to not be present at or before baseline and were verified by the study team. These data are not to be confused with the SAFTEE secondary outcome reporting, which was self reported and not verified nor attributed to the study. The SAE's reported in this table occurred after discontinuing the study medication.
Arm/Group | Riluzole Addition to SSRI Antidepressant | Riluzole/Placebo Addition to SSRI Antidepressant | Placebo Addition to Standard SSRI Antidepressant
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/39 | 2/40
Other Adverse Events (participants affected / at risk) | 19/25 | 31/39 | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole Addition to SSRI Antidepressant (N=25) | Riluzole/Placebo Addition to SSRI Antidepressant (N=39) | Placebo Addition to Standard SSRI Antidepressant (N=40)
Global Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riluzole Addition to SSRI Antidepressant (N=25) | Riluzole/Placebo Addition to SSRI Antidepressant (N=39) | Placebo Addition to Standard SSRI Antidepressant (N=40)
Abdominal Pain (General disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Back Pain (General disorders) | 3 | 3 | 4
Blurred Vision (Eye disorders) | 1 | 0 | 3
Body Aches (General disorders) | 0 | 0 | 2
Bruising (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Clenching Teeth (General disorders) | 0 | 2 | 1
Cold/Flu Symptoms (Infections and infestations) | 3 | 13 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 7 | 6
Dizziness (General disorders) | 0 | 4 | 3
Fall (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 5 | 6 | 8
Frequent Urination (Renal and urinary disorders) | 2 | 2 | 0
GI Issues (Gastrointestinal disorders) | 1 | 3 | 5
Headache (General disorders) | 7 | 11 | 8
Insomnia (General disorders) | 1 | 3 | 2
Leg Pain/Stiffness (General disorders) | 1 | 4 | 3
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Nasal Congestion/Pain (Infections and infestations) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 8 | 11
Nightmares (General disorders) | 1 | 2 | 1
Numbness (Nervous system disorders) | 0 | 2 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Sexual Dysfunction (General disorders) | 1 | 2 | 1
Sleep Disturbance (General disorders) | 2 | 2 | 4
Drowsiness (General disorders) | 1 | 2 | 1
Stomach Pain (Gastrointestinal disorders) | 0 | 2 | 1
Sweating (Nervous system disorders) | 0 | 0 | 2
Tingling Sensation (Nervous system disorders) | 1 | 2 | 1
Toothache (General disorders) | 0 | 0 | 2
Vivid Dreams (General disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes